CLINICAL TRIAL: NCT04335695
Title: Standardized Vascular Rehabilitation Program to Improve Patient Disease and Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not feasible-Not able to enroll the patient population
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019-309
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Vascular Diseases; Peripheral Artery Disease; Peripheral Vascular Diseases
MeSH Terms: conditions — Vascular Diseases; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: All subjects will enroll in the Vascular Rehab program at Baylor Scott & White Heart Hospital and be followed for 1 year after the program ends.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascular Rehabilitation and Follow Up (Other): All subjects will be enrolled in a 6-12 Vascular Rehab Program (VRP) and then be followed for one year following discharge from the VRP.
  Interventions: Behavioral: Vascular Rehabilitation

INTERVENTIONS:
Behavioral: Vascular Rehabilitation — Vascular rehabilitation is a supervised exercise therapy program that includes healthy lifestyle changes to help patients gain strength, energy and confidence to return to daily activities. A program of supervised exercise rehabilitation is considered a primary treatment for people with Peripheral Artery Disease and Intermittent Claudication. In addition, patients will be given a wrist-worn activity tracker and be in contact with a research coordinator every 3 months after they are discharged from the Vascular Rehab program.

SUMMARY:
The purpose of this study is to identify the type of patients being referred for the Vascular Rehabilitation Program (VRP) and to study the success rates of the program according to improvements in walking distance and quality of life surveys. Subjects will be in the VRP for 6-12 weeks and then be followed for 12 months after they complete the program. This is a single-site study at Baylor Scott & White Heart Hospital-Plano.

DETAILED DESCRIPTION:
Peripheral arterial occlusive disease (PAOD) affects 8.5 million people in the United States. One of the most common symptoms of PAOD is claudication. While there are surgical and endovascular treatments to address the underlying arterial occlusions and relieve patients from their symptoms, the initial and primary treatment of vasculogenic claudication is exercise. Numerous studies have documented the success rates of conservative management in the short and long term. However, the main barriers to the use and success of this treatment have been physician reluctance to prescribe and supervise and lack of enthusiasm by the patients. Furthermore, unlike cardiac rehabilitation, supervised rehabilitation and therapy was not a covered benefit for patients until recently.

Beginning in 2018, Centers for Medicare Services (CMS) mandated coverage for supervised therapy for vasculogenic claudication. In 2019, a vascular rehabilitation program was established at The Heart Hospital Plano. As healthcare moves from a fee-for-service model to a payment-for-quality model, treatments such as this are becoming more important. It is necessary to have a better understanding of qualifying patients, the success of this treatment, and the durability and risk factors for success and failure in the real world outside of randomized trials.

This will be the first study of vascular rehabilitation as therapy for vasculogenic claudication in the community setting since this benefit was approved by CMS. It will integrate the areas of Vascular Surgery, Cardiology, Nursing and Cardiac Rehabilitation into a single collaborative project. The project also nicely aligns with the Baylor Scott&White Healthcare System goal of population management in evaluating this lifestyle treatment as an alternative to intervention.

This is a prospective, non-randomized, observational study designed to demonstrate clinically significant benefit in patients undergoing the vascular rehabilitation program at The Heart Hospital Plano.

Informed consent will be obtained from all patients who wish to be enrolled in the study and will be asked to complete quality-of-life surveys specific for vasculogenic claudication (VascuQoL [Appendix 5] and Walking Impairment Questionnaire [Appendix 6]) at their study intake visit, study exit visit, and at 3, 6, 9, and 12 months following discharge from the rehabilitation program. The 3, 6, 9, and 12-month collection periods will be performed via phone.

Ankle brachial indices will be obtained at the time of study enrollment and again at the completion of the rehabilitation program according to standard practice.

A full medical history and relevant demographic and clinical information will be recorded in a de-identified database. This will include but not be limited to age, gender, BMI, tobacco use and medications. Appendix 1.

Walking distance until symptoms occur and total walking distance will be assessed at the study intake and study exit visits and at 3-month intervals for an additional 12 months. Assessments obtained during the 3-month intervals may be obtained via telephone and remote patient monitoring via the activity tracker if possible. Pain scores related to the claudication will be recorded on a scale of 1-4. Appendix 2. Appendix 3.

Every patient will be given a wrist-worn activity tracker to track their daily walking habits during the time period that they are enrolled in the study. This data will be downloaded and stored in the de-identified database.

Following discharge from the vascular rehabilitation program, patients will be contacted every three-months for a year for a follow up quality-of-life survey and walking distance and claudication assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the vascular rehabilitation program at The Heart Hospital Cardiac Rehabilitation Facility.
2. Female or male patients ≥18 years of age.
3. Patient must be accessible for treatment and follow-up.
4. Agrees to wear the activity tracker wrist-worn device
5. Agrees to the follow-up QOL survey schedule
6. Agrees to the follow-up ABI schedule
7. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Declines participation in the study.
2. Has a life-expectancy less than 18 months.
3. Unable to complete necessary study follow-up procedures.
4. Unwilling to wear the wrist-worn activity tracker device.
5. Women who are pregnant.
6. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

   1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
   2. home oxygen
   3. neurologic or orthopedic conditions limiting ability to appropriately comply with rehabilitation program.
   4. class III or class IV NY class congestive heart failure
7. Concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Changes in ankle brachial indices at baseline of VRP and at the termination of VRP (6-12 weeks) (ABI range 0-2) | 6-12 weeks (depending on time in the VRP)
  ABI will be obtained according to standard practice. Severe disease= <=0.4; Mild to moderate disease= 0.41-0.9; Normal= >1.0
Changes to quality of life surveys at VRP enrollment, VRP discharge, and one year after discharge. Range 7-175 | Baseline to 1 year after discharge
  Quality-of-life survey specific for vasculogenic claudication (VascuQoL) (Range QOL not impacted=175; QOL poorly impacted=7)
Changes to walking distance until symptoms of claudication at VRP enrollment, VRP discharge, and at one year post discharge | Baseline to 1 year after discharge
Changes to total walking distance at VRP enrollment, VRP discharge, and at one year post discharge | 13-15 months
  These will be obtained in the VRP at beginning of VRP and termination of VRP. These measurements will also be obtained during the 3-month intervals may be obtained via telephone and remote patient monitoring via the activity tracker if possible. Pain scores related to the claudication will be recorded on a scale of 1-4.

SECONDARY OUTCOMES:
Determination of activity level evaluated on daily, weekly, monthly and cumulative levels | Baseline to 1 year after discharge
  Measurement of activity (walking distance from pedometer)
Rate of lower extremity revascularization intervention that occurs during the study period (1 year following program discharge). | Baseline to 1 year after discharge

CONTACTS AND LOCATIONS:
Overall Officials: William P Shutze, MD, Principal Investigator — Baylor Scott & White Heart Hospital Plano
Locations (1):
- Baylor Scott & White Heart Hospital- Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We don't plan to shared IPD outside our organization but plan to share the cumulative results of the study.

REFERENCES:
- [Background] Malgor RD, Alahdab F, Elraiyah TA, Rizvi AZ, Lane MA, Prokop LJ, Phung OJ, Farah W, Montori VM, Conte MS, Murad MH. A systematic review of treatment of intermittent claudication in the lower extremities. J Vasc Surg. 2015 Mar;61(3 Suppl):54S-73S. doi: 10.1016/j.jvs.2014.12.007. Epub 2015 Feb 23. PMID 25721067
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- [Background] Conijn AP, Jens S, Terwee CB, Breek JC, Koelemay MJ. Assessing the quality of available patient reported outcome measures for intermittent claudication: a systematic review using the COSMIN checklist. Eur J Vasc Endovasc Surg. 2015 Mar;49(3):316-34. doi: 10.1016/j.ejvs.2014.12.002. Epub 2015 Jan 22. PMID 25618453
- [Background] Conijn AP, Loukachov VV, Bipat S, Koelemay MJ. Test-retest Reliability and Measurement Error Are Excellent for the Dutch Version of the VascuQol Questionnaire in Patients with Intermittent Claudication. Eur J Vasc Endovasc Surg. 2015 Oct;50(4):502-5. doi: 10.1016/j.ejvs.2015.07.007. Epub 2015 Aug 8. PMID 26264883
- [Background] Conijn AP, Jonkers W, Rouwet EV, Vahl AC, Reekers JA, Koelemay MJ. Introducing the Concept of the Minimally Important Difference to Determine a Clinically Relevant Change on Patient-Reported Outcome Measures in Patients with Intermittent Claudication. Cardiovasc Intervent Radiol. 2015 Oct;38(5):1112-8. doi: 10.1007/s00270-015-1060-0. Epub 2015 Mar 14. PMID 25772399